CLINICAL TRIAL: NCT05571813
Title: An Open-label, Randomized, Fasted, Single-dose, Three-way Crossover Study to Compare the Pharmacokinetic Characteristics and Safety Between Administration of CKD-341 and Administration of D958 in Healthy Adults
Brief Title: Exploratory Trial to Evaluate the Pharmacokinetic Properties and Safety of CKD-341 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A126_01BE2205P
Record Dates: First submitted 2022-10-06; First posted 2022-10-07 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period1: D958 Period2: CKD-341 Formulation I Period3: CKD-341 Formulation II
  Interventions: Drug: CKD-341
- Sequence 2 (Experimental): Period1: CKD-341 Formulation II Period2: D958 Period3: CKD-341 Formulation I
  Interventions: Drug: CKD-341
- Sequence 3 (Experimental): Period1: CKD-341 Formulation I Period2: CKD-341 Formulation II Period3: D958
  Interventions: Drug: CKD-341
- Sequence 4 (Experimental): Period1: CKD-341 Formulation II Period2: CKD-341 Formulation I Period3: D958
  Interventions: Drug: CKD-341
- Sequence 5 (Experimental): Period1: CKD-341 Formulation I Period2: D958 Period3: CKD-341 Formulation II
  Interventions: Drug: CKD-341
- Sequence 6 (Experimental): Period1: D958 Period2: CKD-341 Formulation II Period3: CKD-341 Formulation I
  Interventions: Drug: CKD-341

INTERVENTIONS:
Drug: CKD-341 — A single dose of 1tablets under fasting condition
  Other Names: D958

SUMMARY:
Exploratory Trial to Evaluate the Pharmacokinetic Properties and Safety of CKD-341 in Healthy Subjects

DETAILED DESCRIPTION:
An open-label, randomized, fasted, single-dose, three-way crossover study to compare the pharmacokinetic characteristics and safety between administration of CKD-341 and administration of D958 in healthy adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, aged ≥ 19 years old at the time of screening
2. Those with a body mass index (BMI) of 17.5 kg/m2 or more and less than 30.5 kg/m2
3. Those who do not have congenital or chronic diseases and have no pathological symptoms or findings as a result of medical examination
4. Clinical laboratory tests (hematology tests, blood chemistry tests, urinalysis, serological tests, etc.) conducted by the principal investigator(or the investigator who has been delegated) according to the characteristics of the drug and screening tests such as vital signs and electrocardiogram tests Result Those who are judged to be suitable as test subjects
5. Before participating in the trial, the purpose and contents of the trial were fully explained, and the participants agreed to participate in this study voluntarily who signed
6. After the first administration of the clinical trial drug, for up to 14 days after the last administration of the investigational drug, you, your spouse, or your partner must agree to maintain the use of an appropriate medically acceptable method of contraception* except for hormonal contraceptives and not donate sperm or eggs ruler
7. Those who have the ability and willingness to participate during the entire examination period

Exclusion Criteria:

1. A history of clinically significant blood, renal, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, psychiatric, neurological, or immune disease (except for simple dental history of calculus, impacted teeth, wisdom teeth, etc.) or evidence one who has 1-1. Patients with hypersensitivity or a history of hypersensitivity to this drug or ingredients contained in this drug, dihydropyridine derivatives, thiazide diuretics, or sulfonamide drugs 1-2. Pregnant (2nd and 3rd trimester) or women who may be pregnant 1-3. Lactating women 1-4. Patients with biliary atresia 1-5. Patient with Severely liver dysfunction 1-6. Patient with Severely aortic valvular stenosis 1-7. Shock patient 1-8. Patients with genetic problems such as intolerance to this drug's additives 1-9. Patients with diabetes or moderate to severe renal impairment (glomerular filtration rate <60mL/min/1.73m2) who used aliskiren-containing agents in combination 1-10. Patients with anuria 1-11. Patients with severe renal failure (creatinine clearance <30 mL/min) 1-12. Patients with refractory hypokalemia 1-13. Patients with hyponatremia and hypercalcemia 1-14. Patients with symptomatic hyperuricemia (history of gout or urolithiasis) 1-15. Untreated Addison's syndrome patients 1-16. Patients receiving lithium therapy 1-17. Patients taking terfenadine or astemizole
2. Those with a history of gastrointestinal diseases (esophageal diseases such as achalasia or esophageal stricture, Crohn's disease) or surgery(except simple appendicectomy, hernia surgery, and tooth extraction surgery) that may affect drug absorption ruler
3. A person who shows the following values as a result of conducting a clinical laboratory test

   - ALT or AST > 2 times the upper limit of the normal range
4. Smokers who smoked more than 20 cigarettes a day within 6 months of screening
5. Those who have taken other clinical investigational drugs or bioequivalence investigational drugs within 6 months before the first administration of the clinical investigational drug
6. Those who meet the following as a result of measuring vital signs at screening

   * Those who have a systolic blood pressure of less than 90 mmHg or more than 140 mmHg or a diastolic blood pressure of less than 60 mmHg or more than 90 mmHg in the sitting position
   * Severe bradycardia (less than 50 beats/min)
7. Those with a history of regular alcohol intake within 1 month of screening

   * More than 14 drinks/Week for women
   * More than 21 drinks/Week for men
8. A person who has taken a drug known to significantly induce or inhibit drug metabolizing enzymes within 30 days before the first administration of the clinical trial drug
9. Those who have taken prescription or non-prescription drugs within 10days prior to the first administration of clinical trial drugs
10. Those who have donated whole blood within 2 months before the first administration of the clinical trial drug, donated component blood within 1 month, received blood transfusion within 1 month, or have plans for the trial during the clinical trial period
11. Those who are judged by the principal investigator (or the person in charge of the test who has been delegated) for reasons other than the above selection/exclusion criteria and are judged unsuitable for participation in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-341, D958 | Pre-dose(0 hour), post-dose 0.25, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72 hours
  Area under the CKD-341, D958 concentration in blood-time curve from zero to final
Cmax of CKD-341, D958 | Pre-dose(0 hour), post-dose 0.25, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72 hours
  The maximum CKD-341, D958 concentration in blood sampling time

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Gyeonggi-do, South Korea